CLINICAL TRIAL: NCT05041426
Title: An Open-label Pilot Protocol to Evaluate the Efficacy of Letermovir for the Prevention of Human Cytomegalovirus (CMV) Infection and Disease in Adult Lung Transplant Recipients With Idiopathic Pulmonary Fibrosis
Brief Title: Letermovir for CMV Prevention After Lung Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fernanda P Silveira, MD, MS (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Fernanda P Silveira, MD, MS, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY21040074
Record Dates: First submitted 2021-04-20; First posted 2021-09-13 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Lung Transplant; CMV
Keywords: Lung transplant; CMV; Letermovir
MeSH Terms: interventions — letermovir; Valganciclovir

STUDY DESIGN:
Intervention Model Description: Interventional, open-label, single center, pilot study with historical controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letermovir (Experimental): Participants who are CMV seropositive (CMV R+) will receive letermovir prophylaxis for 6 months, and participants who are CMV donor seropositive/recipient seronegative (CMV D+/R-) will receive letermovir prophylaxis for 12 months. Letermovir will be administered at a dose of 480 mg IV or oral once daily. IV administration will occur only for those patients unable to swallow tablets. If letermovir is co-administered with cyclosporine A, the dosage of letermovir will be decreased to 240 mg once daily.
  Interventions: Drug: Letermovir
- Valganciclovir (Active Comparator): Historical controls will be lung transplant recipients for idiopathic pulmonary fibrosis from 2010-2019 who are CMV R+ or CMV D+/R-. CMV prophylaxis in the historical controls was with valganciclovir for 6 months for CMV R+ and for 12 months for CMV D+/R-.
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Letermovir — Participants who are CMV R+ will receive LET prophylaxis for 6 months, and participants who are CMV D+/R- will receive LET prophylaxis for 12 months. The duration of prophylaxis is per current standard of care. LET will be administered at a dose of 480 mg IV or oral once daily. IV administration will occur only for those patients unable to swallow tablets. If LET is co-administered with cyclosporin A (CsA), the dosage of LET should be decreased to 240 mg once daily. All patients will be followed for 12 weeks after completion of LET for the occurrence of CMV infection or disease after prophylaxis. Participants on this protocol will receive acyclovir 400 mg orally BID for the duration of LET therapy for herpes simplex virus and varicella zoster virus prophylaxis.
  Other Names: Prevymis
  Arms: Letermovir
Drug: Valganciclovir — Historical controls will have received CMV prophylaxis with valganciclovir for 6 months for CMV R+ and for 12 months for CMV D+/R-.
  Arms: Valganciclovir

SUMMARY:
This is an interventional, open-label, single center, pilot study with historical controls to test the efficacy of letermovir (LET) for the prevention of CMV infection and disease in adult lung transplant recipients (LTRs) with idiopathic pulmonary fibrosis (IPF).

DETAILED DESCRIPTION:
Approximately 30 patients with IPF listed for lung transplantation will be enrolled and 15 are expected to undergo lung transplantation during the study period and receive the intervention. Patients who are CMV seropositive will receive letermovir for 6 months, patients who are CMV seronegative and receive lungs from a CMV seropositive donor (CMV D+/R-) will receive letermovir for 12 months. All patients will be followed for 12 weeks after completion of letermovir for the occurrence of CMV infection or disease after prophylaxis.

Historical controls will be LTRs for IPF from 2010-2019 who are CMV R+ or CMV D+/R- (donor positive/recipient negative). CMV prophylaxis in the historical controls was with valganciclovir for 6 months for CMV R+ and for 12 months for CMV D+/R-. Patients will be matched for CMV serostatus, induction immunosuppression, age, and telomere length.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years on day of signing informed consent
* Listed for lung transplantation (single or double) due to a diagnosis of IPF or receipt of a lung transplant (single or double) for IPF in the 72 hours prior to enrollment
* Have a documented positive serostatus for CMV (CMV IgG seropositive, R+)
* Have a documented negative serostatus for CMV (CMV IgG seronegative, R-) and anticipate receiving or having received a lung allograft from a CMV IgG positive donor, D+). Only participants who are R+ or who are CMV D+/R- will receive intervention. Participants who are CMV D-/R- will be considered screen failures
* Able to travel to UPMC for routine post-transplant visits for a minimum of 15 months after transplantation
* Able to provide informed consent
* Be willing to use a contraceptive method while receiving LET and for at least 90 days following last dose of LET

Exclusion Criteria:

* Receipt of a previous solid organ transplant or hematopoietic stem cell transplant
* Multi-organ transplant recipient, i.e., heart-lung or lung-liver
* HIV seropositive
* HCV antibody or HCV RNA positive
* Donor HCV NAT positive
* Anticipated need for use of ganciclovir, valganciclovir, foscarnet, or cidofovir at the time of transplant
* Known or suspected hypersensitivity to LET or acyclovir
* CrCl < 10 ml/min or dialysis on day of transplant
* Child-Pugh Class C severe hepatic insufficiency
* Pregnancy or expected to conceive while on LET and through at least 90 days following cessation of LET

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of CMV infection or disease during prophylaxis | 6-12 months post-transplant
  Proportion of lung transplant recipients with idiopathic pulmonary fibrosis with CMV infection or disease during letermovir prophylaxis. This will be compared to the proportion of CMV infection or disease in historical lung transplant recipients with idiopathic pulmonary fibrosis who received valganciclovir prophylaxis
Occurrence of CMV infection or disease in the 3 months following completion of prophylaxis | 12 weeks after completion of letermovir
  Proportion of lung transplant recipients with idiopathic pulmonary fibrosis with CMV infection or disease in the 3 months following completion of prophylaxis with letermovir. This will be compared to the proportion of CMV infection or disease in the 3 months following in historical lung transplant recipients with idiopathic pulmonary fibrosis who received valganciclovir prophylaxis.

SECONDARY OUTCOMES:
Discontinuation events | 6-12 months
  Discontinuation of letermovir will be compared to discontinuation of valganciclovir in historical controls
Occurrence of leukopenia or neutropenia while on prophylaxis | 6-12 months
  Proportion of participants who develop any of the following while receiving letermovir: total WBC count ≤ 3,500 cells/mL or absolute neutrophil count ≤ 1,000 cells/mL. This will be compared to the rate of total WBC count ≤ 3,500 cells/mL or absolute neutrophil count ≤ 1,000 cells/mL in historical controls while receiving valganciclovir prophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Silveira, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data outside of our investigative team. Aggregate data will be shared in publications as appropriate.